CLINICAL TRIAL: NCT06975813
Title: Efficacy of Isolated Masseter Versus Masseter- Sternocleidomastoid Trigger Points Injection by Magnesium Sulfate for Myofacial Pain
Brief Title: Magnesium Sulfate and Trigger Points
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, associate professor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- masseter muscle (Active Comparator)
  Interventions: Drug: masseter muscle
- masseter and sternocleidomastoid muscles (Experimental)
  Interventions: Drug: masseter and sternocleidomastoid muscle

INTERVENTIONS:
Drug: masseter muscle — masseter muscle trigger points injection by magnesium sulphate
  Arms: masseter muscle
Drug: masseter and sternocleidomastoid muscle — masseter and sternocleidomastoid muscle trigger points injection by magnesium sulphate
  Arms: masseter and sternocleidomastoid muscles

SUMMARY:
The patients will be randomly assigned to one of the two groups according to the treatment method: group I (masseter group) and group II (masseter &sternocleidomastoid group) where each patient will be injected 0.5ml in each trigger point (TrPs) of magnesium sulphate according to the treatment group by the same operator. The treatment method for TrPs will be the primary predictor variable. Patients will be examined at the following intervals: during diagnosis, 1-month, 3-months, and 6-months post-injection. The participated patients will be assessed using pain score measured on a 10-point visual analogue scale (VAS), the 0 indicating no pain and 10 indicating the worst pain ever

ELIGIBILITY:
Inclusion Criteria:

* definite diagnosis of myofascial pain
* presence of one or more unilateral or bilateral trigger points in the masseter muscle and sternocleidomastoid muscle;
* no history of any invasive procedures of the related masseter muscle.

Exclusion Criteria:

* any painful conditions (other than myofascial trigger points) affecting the orofacial region
* any systemic diseases that could masticatory function (e.g., rheumatoid arthritis and epilepsy);
* pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
muscle pain | 6 months
  by visual analogue scal